CLINICAL TRIAL: NCT05222204
Title: Intraperitoneal (IP) Cisplatin Combined With Intravenous Gemcitabine + Nab-paclitaxel in Patients With Pancreatic Cancer With Peritoneal Metastasis
Brief Title: DDP ip Combined With AG in PDAC With Peritoneal Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-38
Record Dates: First submitted 2021-09-14; First posted 2022-02-03 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Infusions, Parenteral; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: two cohort: cohort A (first-line) and cohort B (post-line with malignant ascites )
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IP (Experimental): intravenous AG+ IP cisplatin
  Interventions: Drug: intraperitoneal (IP) Cisplatin combined with intravenous gemcitabine + nab-paclitaxel

INTERVENTIONS:
Drug: intraperitoneal (IP) Cisplatin combined with intravenous gemcitabine + nab-paclitaxel — intraperitoneal (IP) Cisplatin combined with intravenous gemcitabine + nab-paclitaxel in patients with pancreatic cancer with peritoneal metastasis

SUMMARY:
intraperitoneal (IP) Cisplatin combined with intravenous gemcitabine + nab-paclitaxel in patients with pancreatic cancer with peritoneal metastasis

ELIGIBILITY:
Inclusion Criteria:

cohort A

Patients should meet the following criteria before treatment to be included in the trial:

1. Voluntarily participate and sign the informed consent;
2. Age ≥18 years old and ≤75 years old, gender is not limited;
3. ECOG score ≤2 points;
4. Pathological diagnosis of pancreatic adenocarcinoma;
5. Advanced pancreatic cancer with intra-abdominal metastasis in imaging assessment, or intra-operative intra-operative findings of intra-abdominal metastasis;
6. The time from the end of adjuvant chemotherapy after surgery is more than 6 months, or they have not received any form of anti-tumor therapy before, including interventional chemoembolization, ablation, radiotherapy, chemotherapy, and molecular targeted therapy;
7. No serious abnormal blood system, heart, lung function and immune deficiency (refer to their respective standards);
8. Blood routine indicators: white blood cells ≥3 × 109/L; absolute neutrophil count ≥1.5 × 109/L; platelets ≥100 × 109/L; hemoglobin ≥9 g/dL;
9. Blood biochemical indexes: AST (SGOT), ALT (SGPT) ≤ 2.5 × upper limit of normal (ULN); total bilirubin (TBIL) ≤ ULN; serum creatinine (CRE) ≤ 1.5 × ULN;
10. Coagulation function: prothrombin time (PT), international normalized ratio (INR) ≤ 1.5 × ULN;
11. Able to comply with research visit plans and other protocol requirements.

inclusion criteria (Cohort B)

Patients should meet the following criteria before treatment to be included in the trial:

1. Voluntarily participate and sign the informed consent;
2. Age ≥18 years old and ≤75 years old, gender is not limited;
3. ECOG score ≤2 points;
4. Pathological diagnosis of pancreatic adenocarcinoma;
5. malignant ascites with positive peritoneal cytology or Laparoscopic exploration processed.
6. At least one systemic chemotherapy has been used;
7. No serious abnormal blood system, heart, lung function and immune deficiency (refer to their respective standards);
8. Blood routine indicators: white blood cells ≥3 × 109/L; absolute neutrophil count ≥1.5 × 109/L; platelets ≥100 × 109/L; hemoglobin ≥9 g/dL;
9. Blood biochemical indexes: AST (SGOT), ALT (SGPT) ≤ 2.5 × upper limit of normal (ULN); total bilirubin (TBIL) ≤ ULN; serum creatinine (CRE) ≤ 1.5 × ULN;
10. Coagulation function: prothrombin time (PT), international normalized ratio (INR) ≤ 1.5 × ULN;
11. Able to comply with research visit plans and other protocol requirements.

Exclusion Criteria:

Patients were excluded from the study if they met any of the following criteria:

1. Associated with other systemic malignant tumors;
2. Single kidney, deformed kidney or poor renal compensation;
3. Have used any other study drug within 7 days before chemotherapy;
4. Patients with central nervous system disease, mental illness, unstable angina pectoris, congestive heart failure, severe arrhythmia and other serious diseases that cannot be controlled;
5. There is a history of allergy to the study drug or drugs of similar structure;
6. Patients who are using and require long-term use of warfarin anticoagulation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  patients the time from enrollment to death from any cause

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
intravenous Gemcitabine+ Nab-paclitaxel combined with IP cisplatin in patients with PDAC with peritoneal metastasis
Supporting Information: Study Protocol